CLINICAL TRIAL: NCT05396222
Title: A Prospective Study of the Safety and Efficacy of 3D-printed Custom-made Non-rigid Biomimetic Implant for Anterior Column Reconstruction in Cervical and Thoracolumbar Spine
Brief Title: A Prospective Study of the Safety and Efficacy of 3D-printed Non-rigid Biomimetic Implant in Cervical and Thoracolumbar Spine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202202015DIPC
Record Dates: First submitted 2022-05-04; First posted 2022-05-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Tumor
Keywords: Spinal Tumor; Reconstruction
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D-printed (Experimental): We developed a 3D printed, custom-made, biomimetic prosthesis, with non-rigid structure, which has been tested in biomechanical study and porcine model, showing good bone formation and less stiffness as well. Therefore, we proposed a prospective clinical study to investigate safety, subsidence, and fusion of this prosthesis.
  Interventions: Device: 3D-printed custom-made non-rigid biomimetic implant

INTERVENTIONS:
Device: 3D-printed custom-made non-rigid biomimetic implant — We developed a 3D printed, custom-made, biomimetic prosthesis, with non-rigid structure, which has been tested in biomechanical study and porcine model, showing good bone formation and less stiffness as well. Therefore, we proposed a prospective clinical study to investigate safety, subsidence, and fusion of this prosthesis.

SUMMARY:
Vertebral body resection is a wide accepted procedure in tumor resection, deformity correction, and anterior decompression in spondylosis, ossification of posterior longitudinal ligaments, and spondylodiscitis surgery. However, reconstruction of segmental defect is still challenging to spine surgeon, especially in 3-column resection, such as total en bloc spondylectomy in tumor patients. Various graft or prosthesis for reconstruction has been reported, such as structural allograft, Harms mesh cages, expandable cages, and carbon fiber stackable cages. There are no high evidence level study examining the superiority of those different methods.

Recently, 3D printed vertebral body replacement has been reported in different disease entities as well, such as tumor, Kümmell's disease in osteoporosis, and spondylosis. 3D printed implant comes with superiority in production of complex geometries and regularity of the fine surface detailed that promote bone ingrowth. Although, 3D-printed titanium vertebra could achieved bone integration in human, a systemic review showed that the subsidence noted in 31.4% of spine surgery with 3D printed implants. In spine surgery, the fixation construct is sufficiently stiff, interbody motion can be reduced, and loading sharing promotes bone fusion. On the other hand, if the reconstruction is too stiff, stress shielding at fusion site occurs. The concept of dynamic fusion, as opposed to rigid fusion, has been demonstrated by an anterior cervical interbody fusion study in porcine model, demonstrating good bone formation, less postfusion stiffness, and a trend to less subsidence.

Thus, we developed a 3D printed, custom-made, biomimetic prosthesis, with non-rigid structure, which has been tested in biomechanical study and porcine model, showing good bone formation and less stiffness as well. Therefore, we proposed a prospective clinical study to investigate safety, subsidence, and fusion of this prosthesis.

DETAILED DESCRIPTION:
This is a single-arm prospective observational phase I clinical study to investigate the safety of the non-rigid 3D printed custom-made biomimetic implant. The implants are made of Titanium alloy. Patient receiving 1- to 3-level corpectomy at cervical and thoracolumbar spine. At first stage, we plan to enroll 3 cervical patients, and 3 thoracolumbar patients with non-rigid 3D printed custom-made biomimetic reconstructions. After 3 months observation after the last patients enrolled, we will conduct an interim investigation to investigate those 6 patients. if there is no re-operations due to acute post-operative reconstruction failure. We will continue the study. Total 9 cervical patients, and 9 thoracolumbar patients will be enrolled. Patients are evaluated preoperatively, right after surgery, and 1, 3, 6, 12 months postoperatively. Measure outcomes included overall success, VAS neck and back pain, patient satisfaction, anxiety score, SF-12 MCS/PCS, complications, subsequent surgery rate, and subsidence and fusion rate on radiological examination. Radiological evaluation, including X-ray and computed tomography, will be done pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively. In addition, neck disability index (NDI) will be evaluated in cervical patents, and SORGSQ 2.0 self-reported questionnaire will be applied for all oncology patients. The primary endpoint was a FDA composite definition of success comprising clinical improvement and absence of major complications and secondary surgery events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 79 years;
2. Patient meet the indication for 1- to 3- level corpectomy, for primary bone tumor at spine, or metastatic tumor at spine.
3. Deficit confirmed by CT, MRI, and X-ray;
4. Pathology level located from C3 to L5.
5. Physically and mentally able and willing to comply with the protocol;
6. Signed informed consent;
7. NTU Spine Multidisciplinary Board confirmed tumor excision surgery is indicated.
8. Life expectancy longer than 6 months (Tokuhashi Scoring System)

Exclusion Criteria:

1. Patient does not meet the indication of corpectomy, which is under the surveillance.
2. More than three vertebrae required corpectomy;
3. Corpectomy levels above C3 and below L5
4. T-score less than -2.5
5. Known allergy to device materials - such as titanium
6. Any diseases or conditions that would preclude accurate clinical evaluation;
7. Daily, high-dose oral and/or inhaled steroid or a history of chronic use of high dose steroids;
8. BMI > 35
9. Life expectancy less than 6 months - (Tokuhashi Scoring System)
10. The subject has received radiation therapy or chemotherapy at the trial site within one year;
11. Anterior spine surgery has been received at or near the spine surgery site;
12. The subject has systemic infection,or focal vertebral infection or trauma;
13. The subject has endocrine disorders or metabolic disorders known to affect bone formation, such as: Paget's disease, renal osteodystrophy, hypothyroidism;
14. The subject has neuromuscular diseases, those at risk of instability, implant fixation failure or postoperative care complications, including: spina bifida, cerebral palsy, and multiple sclerosis;
15. Osteopenia, osteomyelitis;
16. Pregnant women.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Patient were evaluated at 12 months postoperatively.
  We will follow up the condition of participants with treatment-related adverse events as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Degree of change in the subsidence | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  In a medical sense, subsidence refers to the collapse or settling of bone located immediately next to an implantable device in direction of the loading force. It is uasually recorded in millimeters. It was assessed on radiological examination. Radiological evaluation, including X-ray and computed tomography.
The percentage of patients with successful fusion | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  The fusion rate is the percentage of patients with successful fusion over a specific range of follow up. The outcomes about fusion rate of bone was assessed on radiological examination. Radiological evaluation, including X-ray and computed tomography.
Pain score | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  Pain score was assessed by Visual Analogue Scale. (0 means no pain, while 10 is the most painful situation).
Short form-12 mental component score | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  The minimum value of mental component scale (MCS-12) is 18.7, and the maximum value of MCS-12 is 65.2. Higher scores mean a better outcome.
Anxiety score | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  Anxiety score was assessed by Beck Anxiety Inventory (The minimum value is 0 and the maximum value is 63. A higher score means a worse outcome).
Neck Disability Index (NDI) | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  Physical function was assessed by Neck Disability Index (NDI), it will be evaluated only in cervical patents.
  An improvement in Neck Disability Index (NDI) score of at least 30 points for a patient with a preoperative NDI score of 60 or greater; or an improvement of at least 50% of preoperative NDI score for patients with a preoperative score of less than 60.
Patient Satisfaction Questionnaire | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  Patients will be surveyed by Patient Satisfaction Questionnaire. There are two questions on the questionnaire to evaluate if they are satisfied with their treatment and if they will recommend their respective surgery to a friend.
Short form-12 physical component score | Patient were evaluated pre-operatively, immediately after the surgery, and 1, 3, 6, 12 months postoperatively.
  The minimum value of physical component scale (PCS-12) is 18.4 and the maximum value of PCS-12 is 57.8.

CONTACTS AND LOCATIONS:
Overall Officials: Fon-Yih Fon-Yih, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Bridwell KH, Lenke LG, McEnery KW, Baldus C, Blanke K. Anterior fresh frozen structural allografts in the thoracic and lumbar spine. Do they work if combined with posterior fusion and instrumentation in adult patients with kyphosis or anterior column defects? Spine (Phila Pa 1976). 1995 Jun 15;20(12):1410-8. PMID 7676341
- [Result] Lewandrowski KU, Hecht AC, DeLaney TF, Chapman PA, Hornicek FJ, Pedlow FX. Anterior spinal arthrodesis with structural cortical allografts and instrumentation for spine tumor surgery. Spine (Phila Pa 1976). 2004 May 15;29(10):1150-8; discussion 1159. doi: 10.1097/00007632-200405150-00019. PMID 15131446
- [Result] Dvorak MF, Kwon BK, Fisher CG, Eiserloh HL 3rd, Boyd M, Wing PC. Effectiveness of titanium mesh cylindrical cages in anterior column reconstruction after thoracic and lumbar vertebral body resection. Spine (Phila Pa 1976). 2003 May 1;28(9):902-8. doi: 10.1097/01.BRS.0000058712.88053.13. PMID 12942006
- [Result] Viswanathan A, Abd-El-Barr MM, Doppenberg E, Suki D, Gokaslan Z, Mendel E, Rao G, Rhines LD. Initial experience with the use of an expandable titanium cage as a vertebral body replacement in patients with tumors of the spinal column: a report of 95 patients. Eur Spine J. 2012 Jan;21(1):84-92. doi: 10.1007/s00586-011-1882-7. Epub 2011 Jun 18. PMID 21681631
- [Result] Boriani S, Biagini R, Bandiera S, Gasbarrini A, De Iure F. Reconstruction of the anterior column of the thoracic and lumbar spine with a carbon fiber stackable cage system. Orthopedics. 2002 Jan;25(1):37-42. doi: 10.3928/0147-7447-20020101-14. PMID 11811240
- [Result] Xu N, Wei F, Liu X, Jiang L, Cai H, Li Z, Yu M, Wu F, Liu Z. Reconstruction of the Upper Cervical Spine Using a Personalized 3D-Printed Vertebral Body in an Adolescent With Ewing Sarcoma. Spine (Phila Pa 1976). 2016 Jan;41(1):E50-4. doi: 10.1097/BRS.0000000000001179. PMID 26335676
- [Result] Glennie RA, Rampersaud YR, Boriani S, Reynolds JJ, Williams R, Gokaslan ZL, Schmidt MH, Varga PP, Fisher CG. A Systematic Review With Consensus Expert Opinion of Best Reconstructive Techniques After Osseous En Bloc Spinal Column Tumor Resection. Spine (Phila Pa 1976). 2016 Oct 15;41 Suppl 20:S205-S211. doi: 10.1097/BRS.0000000000001835. PMID 27488296
- [Result] Choy WJ, Mobbs RJ, Wilcox B, Phan S, Phan K, Sutterlin CE 3rd. Reconstruction of Thoracic Spine Using a Personalized 3D-Printed Vertebral Body in Adolescent with T9 Primary Bone Tumor. World Neurosurg. 2017 Sep;105:1032.e13-1032.e17. doi: 10.1016/j.wneu.2017.05.133. Epub 2017 May 31. PMID 28578109
- [Result] Wei F, Li Z, Liu Z, Liu X, Jiang L, Yu M, Xu N, Wu F, Dang L, Zhou H, Li Z, Cai H. Upper cervical spine reconstruction using customized 3D-printed vertebral body in 9 patients with primary tumors involving C2. Ann Transl Med. 2020 Mar;8(6):332. doi: 10.21037/atm.2020.03.32. PMID 32355776
- [Result] Yang X, Wan W, Gong H, Xiao J. Application of Individualized 3D-Printed Artificial Vertebral Body for Cervicothoracic Reconstruction in a Six-Level Recurrent Chordoma. Turk Neurosurg. 2020;30(1):149-155. doi: 10.5137/1019-5149.JTN.25296-18.2. PMID 31049920
- [Result] Girolami M, Boriani S, Bandiera S, Barbanti-Brodano G, Ghermandi R, Terzi S, Tedesco G, Evangelisti G, Pipola V, Gasbarrini A. Biomimetic 3D-printed custom-made prosthesis for anterior column reconstruction in the thoracolumbar spine: a tailored option following en bloc resection for spinal tumors : Preliminary results on a case-series of 13 patients. Eur Spine J. 2018 Dec;27(12):3073-3083. doi: 10.1007/s00586-018-5708-8. Epub 2018 Jul 23. PMID 30039254
- [Result] Dong C, Wei H, Zhu Y, Zhou J, Ma H. Application of Titanium Alloy 3D-Printed Artificial Vertebral Body for Stage III Kummell's Disease Complicated by Neurological Deficits. Clin Interv Aging. 2020 Dec 2;15:2265-2276. doi: 10.2147/CIA.S283809. eCollection 2020. PMID 33293803
- [Result] Wei F, Xu N, Li Z, Cai H, Zhou F, Yang J, Yu M, Liu X, Sun Y, Zhang K, Pan S, Wu F, Liu Z. A prospective randomized cohort study on 3D-printed artificial vertebral body in single-level anterior cervical corpectomy for cervical spondylotic myelopathy. Ann Transl Med. 2020 Sep;8(17):1070. doi: 10.21037/atm-19-4719. PMID 33145289
- [Result] Fang T, Zhang M, Yan J, Zhao J, Pan W, Wang X, Zhou Q. Comparative Analysis of 3D-Printed Artificial Vertebral Body Versus Titanium Mesh Cage in Repairing Bone Defects Following Single-Level Anterior Cervical Corpectomy and Fusion. Med Sci Monit. 2021 Feb 7;27:e928022. doi: 10.12659/MSM.928022. PMID 33550326
- [Result] Girolami M, Sartori M, Monopoli-Forleo D, Ghermandi R, Tedesco G, Evangelisti G, Pipola V, Pesce E, Falzetti L, Fini M, Gasbarrini A. Histological examination of a retrieved custom-made 3D-printed titanium vertebra : Do the fine details obtained by additive manufacturing really promote osteointegration? Eur Spine J. 2021 Oct;30(10):2775-2781. doi: 10.1007/s00586-021-06926-w. Epub 2021 Jul 16. PMID 34279722
- [Result] Wallace N, Schaffer NE, Aleem IS, Patel R. 3D-printed Patient-specific Spine Implants: A Systematic Review. Clin Spine Surg. 2020 Dec;33(10):400-407. doi: 10.1097/BSD.0000000000001026. PMID 32554986
- [Result] Yang SH, Xiao FR, Lai DM, Wei CK, Tsuang FY. A Dynamic Interbody Cage Improves Bone Formation in Anterior Cervical Surgery: A Porcine Biomechanical Study. Clin Orthop Relat Res. 2021 Nov 1;479(11):2547-2558. doi: 10.1097/CORR.0000000000001894. PMID 34343157